CLINICAL TRIAL: NCT00891111
Title: Incentives for Preventative Health Care: Increasing Completion of Health Risk Assessments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carnegie Mellon University (Other)
Collaborators: Yale University (Other); University of Pennsylvania (Other)
Responsible Party: Principal Investigator, George Loewenstein, Professor, Carnegie Mellon University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CMUHS08613
Record Dates: First submitted 2009-04-30; First posted 2009-05-01 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Prevention
Keywords: Health Risk Assessment; Incentives; Preventative Healthcare; Encouraging Health Risk Assessments

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Direct Payment (Experimental): Direct Payment: Employees receive a $25 gift card upon completion of a Health Risk Assessment
  Interventions: Behavioral: Direct Payment
- Regret Lottery (Experimental): Regret Lottery: Employees are divided into work units of about 5 employees. Employees in the lottery-linked incentive condition will be eligible for a weekly lottery drawing only if they have already completed their health risk assessment. The lotteries will work as follows. Participants will be assigned to work units of about 10 people. Each week, one work group is drawn at random. If a participants group was drawn and that participant already completed the health risk assessment, then that person will win a $100 cash prize. If all of the members of his or her work group also filled out the health risk assessment, then the prize will be boosted.
  Interventions: Behavioral: Regret Lottery

INTERVENTIONS:
Behavioral: Direct Payment — $25 gift card given upon completion of Health Risk Assessment
  Arms: Direct Payment
Behavioral: Regret Lottery — Entered into a lottery upon completion of Health Risk Assessment
  Arms: Regret Lottery

SUMMARY:
The purpose of this study is to understand using incentives to encourage employees to increase participation in an aspect of a corporate wellness program - filling out health risk assessments. This study will test whether lottery-linked incentives are more effective than guaranteed incentives in encouraging people to fill out health risk assessments.

This study will be run in an employer setting in which rates of health risk assessment completion are suboptimal. This study would be conducted within a workplace setting in which the firm is divided into a number of geographically situated and functionally related subunits. The investigators will run a "complete your health risk assessment now!" program for 4 weeks. Each work unit will obtain a symbol. Every week, one symbol will be randomly drawn, publicly announced, and anyone in that work unit at the firm who has received their preventive screening would receive a $100 prize. In addition, if all of employees in that unit have completed their forms, then the prize will be increased to $125.

The investigators expect this condition to result in greater compliance compared to a control condition in which employees would receive weekly reminders and a direct payment of a $25 gift card for completing the form at anytime during the 4 weeks of the study. This is analogous to direct payments that have been used by insurers to encourage completion of such forms in other contexts.

DETAILED DESCRIPTION:
The purpose of this study is to apply concepts from behavioral economics to increase the effectiveness of incentives for preventative health care.

Health risk assessments are an important part of preventative healthcare. Employees fill out these forms and are given feedback about their health risks and steps they can take to improve their health. This study will be run in an employer setting in which rates of health risk assessment completion are suboptimal. This study would be conducted within a workplace setting in which the firm is divided into a number of geographically situated and functionally related subunits. We will run a "complete your health risk assessment now!" program for 4 weeks. Each work unit will obtain a symbol. Every week, one symbol will be randomly drawn, publicly announced, and anyone in that work unit at the firm who has received their preventive screening would receive a $100 prize. In addition, if all of employees in that unit have completed their forms, then the prize will be increased to $125.

This program plays on a number of psychological factors: 1) avoidance of regret, which one will experience if the number/symbol of the unit one is a member of is drawn and one does not win a prize because one is not participating in the wellness program 2) amplification of such regret by social means - because other people around you who are participating will receive cash prizes 3) mild social pressure, because high enrollments will yield benefits for all participants.

ELIGIBILITY:
Inclusion Criteria:

* Full time employees

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 634 (Actual)
Dates: Start 2009-05; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Percent of people in each condition who complete their health risk assessment | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: George Loewenstein, PhD, Principal Investigator — Carnegie Mellon University
Locations (8):
- United States (8):
  - Med3000, Shelton, Connecticut
  - Med 3000, Pensacola, Florida
  - Med3000, Tampa, Florida
  - Med3000, Tinley Park, Illinois
  - Med3000, Winston-Salem, North Carolina
  - Med3000, Dayton, Ohio
  - Med3000, Pittsburgh, Pennsylvania
  - Med3000, Dallas, Texas